CLINICAL TRIAL: NCT06861088
Title: A Randomized, Placebo-Controlled, Double-Blind Phase 3 Trial Comparing, Relative to Placebo, the Effect of Kinisoquin™ on Thromboembolic Events in Patients With Metastatic or Locally Advanced Pancreatic Cancer (CATIQ P3)
Brief Title: The Effect of Kinisoquin™ on Thromboembolic Events in Patients With Metastatic or Locally Advanced Pancreatic Cancer
Acronym: CATIQ P3
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Quercis Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IQC-CAT-301
Expanded Access: Available
Record Dates: First submitted 2025-02-28; First posted 2025-03-06 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Venous Thromboembolism; Metastatic Pancreatic Cancer; Locally Advanced Pancreatic Adenocarcinoma
Keywords: Metastatic Pancreatic Cancer; Pancreatic Adenocarcinoma; Thromboembolism; Cancer-associated Thrombosis; Deep Vein Thrombosis; Pulmonary Embolism; Chemotherapy-associated VTE; Locally Advanced Pancreatic Cancer
MeSH Terms: conditions — Venous Thromboembolism; Pancreatic Neoplasms; Thromboembolism; Venous Thrombosis; Pulmonary Embolism | interventions — isoquercitrin

STUDY DESIGN:
Intervention Model Description: Initially, patients will be randomized on a 1:1:1 basis to Kinisoquin™ 1000 mg, Kinisoquin™ 2000 mg, or matching placebo daily. Kinisoquin™ or placebo will be administered orally at 8 capsules per day for 16 weeks (4 capsules in the morning and 4 capsules in the evening). An interim analysis will be performed when 26 positively adjudicated primary endpoint events have been attained across all three arms, expected to have been accrued after enrolment of the 180th patient.
  Deselected dose patients will be followed long term for progression-free survival and overall survival but will not be included in the final primary endpoint analysis.
  Futility will be assessed at the interim and, if passed, the better performing dose will be identified and a sample size reassessment performed; thereafter, randomization to the study will continue only for the selected dose and placebo on a 1:1 basis.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Kinisoquin™ 1000mg (Experimental): Initially, patients will be randomized on a 1:1:1 basis to Kinisoquin™ 1000mg, Kinisoquin™ 2000mg or matching placebo daily. Patients in the 1,000 mg group will receive Kinisoquin™ at a total daily dose of 1,000 mg, administered orally as two 250 mg Kinisoquin™ capsules and two placebo capsules in the morning, and two 250 mg Kinisoquin™ capsules and two placebo capsules in the evening (total of 8 capsules daily) for 16 weeks.
  An interim analysis will be performed when 26 positively adjudicated primary endpoint events have been attained across all three arms and the best performing dose will be identified and a sample size reassessment performed. Thereafter, randomization to the study will continue only for the selected dose and placebo on a 1:1 basis.
  Interventions: Drug: Kinisoquin™
- Kinisoquin™ 2000mg (Experimental): Initially, patients will be randomized on a 1:1:1 basis to Kinisoquin™ 1000mg, Kinisoquin™ 2000mg or matching placebo daily. Patients in the 2,000 mg group will receive Kinisoquin™ at a total daily dose of 2,000 mg, administered orally as four 250 mg Kinisoquin™ capsules in the morning and four 250 mg Kinisoquin™ capsules in the evening (total of 8 capsules daily) for 16 weeks.
  An interim analysis will be performed when 26 positively adjudicated primary endpoint events have been attained across all three arms and the best performing dose will be identified and a sample size reassessment performed. Thereafter, randomization to the study will continue only for the selected dose and placebo on a 1:1 basis.
  Interventions: Drug: Kinisoquin™
- Placebo (Placebo Comparator): Patients in this group will be administered placebo orally at 8 capsules per day for 16 weeks (4 capsules in the morning and 4 capsules in the evening).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Kinisoquin™ — Kinisoquin™ capsules formulated with vitamin C and vitamin B3
  Other Names: Isoquercetin
  Arms: Kinisoquin™ 1000mg; Kinisoquin™ 2000mg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The aim of this Phase 3 study is to evaluate the efficacy of Kinisoquin™ as compared to the placebo in prevention of thromboembolic events in patients with metastatic or locally advanced pancreatic cancer.

DETAILED DESCRIPTION:
Approximately one-third of all pancreatic cancer patients suffer from a venous thromboembolism (VTE). The greatest risk of thrombosis is observed in the first three months following the start of chemotherapy. The development of distant metastasis in pancreatic cancer increases the risk of VTE approximately 4-fold.

Kinisoquin™ is a more bioavailable form of quercetin, a naturally occurring flavonol, intended to prevent thromboembolic events in cancer patients. The aim of this study is to evaluate the efficacy of Kinisoquin™ in prevention of thromboembolic events in patients with metastatic or locally advanced pancreatic cancer.

This trial is a randomized, placebo-controlled, double-blinded, Phase 3 trial in metastatic or locally advanced pancreatic cancer patients who are initiating chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have histological or cytological confirmed pancreatic adenocarcinoma malignancy that is metastatic (including recurrent with distant metastases) or locally advanced.
2. Receiving first line chemotherapy (within 45 days of first dose of study drug) Note: subjects must be either initiating first systemic cancer therapy regimen following initial diagnosis or initiating first cycle of chemotherapy for disease recurrence.
3. Minimum age 18 years.
4. Life expectancy of greater than 4 months.
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
6. Participants must have preserved organ and marrow function as defined by:

   * Platelet count ≥ 100,000/mcL.
   * Prothrombin time (PT) and partial thromboplastin time (PTT) ≤ 1.5x institutional upper limit of normal (ULN).
   * Total bilirubin ≤ 3x ULN without liver metastases and < 5x ULN in presence of liver metastases.
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3x ULN without liver metastases and < 5x ULN in the presence of liver metastases
   * Estimated creatinine clearance (CrCl > 30 mL/min).
7. Willingness of women of child-bearing potential and men to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation until at least 4 weeks after study completion.
8. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Participants with known brain metastases
2. Prior history of documented thromboembolic event within the last 12 months (excluding central line associated events whereby patients completed anticoagulation)
3. Active bleeding or high risk for bleeding (e.g. known acute gastrointestinal ulcer)
4. History of significant hemorrhage (requiring hospitalization or transfusion) outside of a surgical setting within the last 24 months
5. Familial bleeding diathesis
6. Known diagnosis of disseminated intravascular coagulation (DIC)
7. Currently receiving anticoagulant therapy
8. Current daily use of aspirin (> 100mg daily), Clopidogrel (Plavix), cilostazol (Pletal), aspirin-dipyridamole (Aggrenox) (within 10 days) or considered to use regular use of higher doses of non-steroidal anti-inflammatory agents as determined by the treating physician (e.g. ibuprofen > 800mg daily or equivalent)
9. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
10. Known intolerance to the active ingredient of Kinisoquin™, isoquercetin, nicotinic acid, or ascorbic acid (including known G6PD deficiency)
11. Females of child-bearing potential who are lactating, have a positive pregnancy test at Screening, or are unwilling to use acceptable contraception prior to study entry and for the duration of study participation until at least 4 weeks after study completion.
12. Participation in other clinical trials The study is open to any individual who has a metastatic or locally advanced pancreatic adenocarcinoma malignancy without discrimination based on race, religion, political affiliation, or other criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2025-12-19 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of Kinisoquin™ | 16 weeks
  The time to the first positively adjudicated thromboembolic event (TE) over 16 weeks of treatment in patients treated with Kinisoquin™ compared with placebo.
Effectiveness of Kinisoquin™ | 16 weeks
  The time to the first positively adjudicated proximal or distal lower extremity DVT, any pulmonary embolism, fatal pulmonary embolism diagnosed on autopsy, catheter-related thrombosis, visceral thrombosis or arterial thrombosis. Events will be classified as incidental or symptomatic: incidental TE will be so classified if the imaging was ordered primarily for staging or re-staging or conducted for reasons other than identification of a thrombosis as compared to the placebo.

SECONDARY OUTCOMES:
Risk of TE | 16 weeks
  To assess the risk of TE defined as proximal or distal lower extremity DVT, any pulmonary embolism, fatal pulmonary embolism diagnosed on autopsy, or arterial thrombosis over 16 weeks of treatment in patients treated with Kinisoquin™ compared with placebo.
Catheter-related TEs | 16 weeks
  To assess the risk of catheter-related TEs over 16 weeks after study treatment initiation in patients treated with Kinisoquin™ compared with placebo.
Risk of major hemorrhage | 16 weeks
  To assess the risk of major hemorrhage in patients treated with Kinisoquin™ compared with placebo according to ISTH definition. The criteria for major hemorrhage in non-surgical patients is:
  * Fatal bleeding, and/or
  * Symptomatic bleeding in a critical area or organ such as intracranial, intraspinal, intraocular, retroperitoneal, intra-articular or pericardial, or intramuscular with compartment syndrome, and/or
  * Bleeding causing a fall in hemoglobin level ≥ 2 g/L or
  * Bleeding leading to a transfusion ≥ 2 units of packed red blood cells
Risk of clinically relevant non-major bleeding | 16 weeks
  To assess the risk of clinically relevant non-major bleeding in patients treated with Kinisoquin™ compared with placebo.
Progression-Free Survival (PFS) | 12 months
  Progression-free survival until 12 months after study treatment initiation according to RECIST, as assessed by the site Investigator's review, in patients treated with Kinisoquin™ compared with placebo.
Overall Survival (OS) | 24 Months
  Overall survival until 24 months after study treatment initiation in patients treated with Kinisoquin™ compared with placebo.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Ventura Clinical Trials, Ventura, California
  - Clavis Medical, LLC, Miami Lakes, Florida
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No